CLINICAL TRIAL: NCT00705783
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of an Intramuscular Depot Formulation of Aripiprazole as Maintenance Treatment in Patients With Schizophrenia
Brief Title: Intramuscular Depot Formulation of Aripiprazole as Maintenance Treatment in Patients With Schizophrenia
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-07-246
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; Intramuscular (IM) depot; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole depot (Experimental): Patients received aripiprazole 300 mg or 400 mg depot intramuscularly every 28 days for 52 weeks.
  Interventions: Drug: Aripiprazole depot
- Placebo depot (Placebo Comparator): Patients received placebo intramuscularly every 28 days for 52 weeks.
  Interventions: Drug: Placebo depot

INTERVENTIONS:
Drug: Aripiprazole depot — Aripiprazole depot was supplied in 400 mg lyophilized vials. Patients received aripiprazole 300 mg if they were unable to tolerate aripiprazole 400 mg.
  Other Names: Abilify
  Arms: Aripiprazole depot
Drug: Placebo depot — Placebo depot was supplied in 400 mg lyophilized vials.
  Arms: Placebo depot

SUMMARY:
The purpose of the trial was to evaluate the efficacy, safety, and tolerability of an intramuscular depot formulation of aripiprazole as maintenance treatment in patients with schizophrenia.

The trial was designed into 4 treatment phases. Phase 1 was designed to allow for a patient to be converted from their current antipsychotic treatment to oral non-generic aripiprazole monotherapy (oral conversion phase from 4 to 6 weeks). During Phase 2, the patient was stabilized on oral non-generic aripiprazole monotherapy (oral stabilization phase from a minimum of 4 weeks to a maximum of 12 weeks). Once the patient was stabilized in Phase 2, they entered Phase 3, the single-blind intramuscular (IM) depot aripiprazole stabilization phase. The goal of the phase was to stabilize the patient on the IM depot aripiprazole formulation for a minimum of 12 weeks to a maximum of 36 weeks. When the patient was stabilized, they were eligible to be randomized into the double-blind IM depot maintenance phase (Phase 4). During Phase 4, the patient was assessed for exacerbation of psychotic symptoms and/or impending relapse for up to 52 weeks.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study consisting of a screening phase and 4 treatment phases. Eligibility was determined during a screening phase of 2 to 42 days. Patients receiving oral treatment with an antipsychotic other than non-generic aripiprazole entered Phase 1. Patients with a lapse in aripiprazole or other antipsychotic treatment at the time of study entry ("lapse" defined as > 3 consecutive days without medication) entered directly into Phase 2. During Phase 1 (oral conversion), patients were cross-titrated during weekly visits from other antipsychotics to oral non-generic aripiprazole monotherapy over a minimum of 4 weeks and a maximum of 6 weeks. During Phase 2 (a minimum of 4 weeks and a maximum of 12 weeks in duration), patients were assessed bi-weekly and stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily. After stability criteria were met in Phase 2, patients entered the single-blind aripiprazole intramuscular (IM) depot stabilization phase, Phase 3. In Phase 3, patients were stabilized on aripiprazole IM depot for 12 consecutive weeks. Once the patient met the stability criteria, they were eligible to be randomized into the double-blind phase, Phase 4. Patients were randomized in a 2:1 ratio (aripiprazole IM depot vs placebo IM depot) stratified by region and last aripiprazole IM depot injection dose level in Phase 3. During Phase 4, patients were assessed for impending relapse/exacerbation of psychotic symptoms. If a patient was identified with impending relapse/exacerbation of psychotic symptoms, they were withdrawn from the trial and given the opportunity to enroll into an open-label aripiprazole IM depot trial, 31-08-248. Patients that completed Phase 4 (up to and including Week 52) had the option to enroll into an open-label aripiprazole IM depot trial, 31-08-248 (NCT00731549).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent and/or consent obtained from a legally acceptable representative (as required by the Institutional Review Board/Institutional Ethics Committee [IRB/IEC]), prior to the initiation of any protocol-required procedures.
* Male and female subjects 18 to 60 years of age, inclusive, at time of informed consent.
* Subjects with a current diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition text revision (DSM-IV-TR) criteria and a history of the illness for at least 3 years prior to screening.
* Subjects who, in the investigator's judgment, require chronic treatment with an antipsychotic medication.
* Subjects able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, IM depot injection, discontinuation of prohibited concomitant medications; who can read and understand the written word in order to complete patient-reported outcomes measures; and who can be reliably rated on assessment scales.

Exclusion Criteria:

* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, or amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Subjects with schizophrenia that are considered resistant/refractory to antipsychotic treatment by history or response only to clozapine.
* Subjects with a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's judgment.
* Subjects who currently meet DSM-IV-TR criteria for substance dependence, including alcohol and benzodiazepines, but excluding caffeine and nicotine; or 2 positive drug screens for cocaine.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones; or hypersensitivity to antipsychotic agents.
* Subjects with uncontrolled thyroid function abnormalities.
* Subjects with a history of seizures, neuroleptic malignant syndrome, clinically significant tardive dyskinesia, or other medical condition that would expose them to undue risk or interfere with study assessments.
* Subjects who are involuntary incarcerated.
* Subjects who have used an investigational agent within 30 days of screening or prior participation in a clinical study with aripiprazole IM depot.
* Subjects with clinically significant abnormalities in laboratory test results, vital signs, or ECG results; and subjects hospitalized for more than 30 days in the 90 days prior to Phase 1.
* Subjects who fail to wash-out from prohibited concomitant medications, including the use of CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers, antipsychotics, antidepressants (including monoamine oxidase inhibitors [MAOI}), and mood stabilizers during screening and/or Phase 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 843 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Sanchez, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (101):
- United States (42):
  - Otsuka Investigational Site, Chandler, Arizona
  - Otsuka Investigational Site, Anaheim, California
  - Otsuka Investigational Site, National City, California
  - Otsuka Investigational Site, Oceanside, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site, Santa Ana, California
  - Otsuka Investigational Site, Highlands Ranch, Colorado
  - Otsuka Investigational Site, Norwalk, Connecticut
  - Otsuka Investigational Site, Altamonte Springs, Florida
  - Otsuka Investigational Site, Bradenton, Florida
  - Otsuka Investigational Site, Hollywood, Florida
  - Otsuka Investigational Site, Maitland, Florida
  - Otsuka Investigational Site, Miami, Florida
  - Otsuka Investigational Site, North Miami, Florida
  - Otsuka Investigational Site, Orange City, Florida
  - Otsuka Investigational Site, Tampa, Florida
  - Otsuka Investigational Site, Atlanta, Georgia
  - Otsuka Investigational Site, Hoffman Estates, Illinois
  - Otsuka Investigational Site, Munster, Indiana
  - Otsuka Investigational Site, Baton Rouge, Louisiana
  - Otsuka Investigational Site, Lake Charles, Louisiana
  - Otsuka Investigational Site, New Orleans, Louisiana
  - Otsuka Investigational Site, Columbia, Maryland
  - Otsuka Investigational Site, Flowood, Mississippi
  - Otsuka Investigational Site, St Louis, Missouri
  - Otsuka Investigational Site, North Platte, Nebraska
  - Otsuka Investigational Site, Albuquerque, New Mexico
  - Otsuka Investigational Site, Buffalo, New York
  - Otsuka Investigational Site, Cedarhurst, New York
  - Otsuka Investigational Site, Elmsford, New York
  - Otsuka Investigational Site, Holliswood, New York
  - Otsuka Investigational Site, Jamaica, New York
  - Otsuka Investigational Site, Staten Island, New York
  - Otsuka Investigational Site, Cleveland, Ohio
  - Otsuka Investigational Site, Oklahoma City, Oklahoma
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Memphis, Tennessee
  - Otsuka Investigational Site, Austin, Texas
  - Otsuka Investigational Site, DeSoto, Texas
  - Otsuka Investigational Site, Bellevue, Washington
  - Otsuka Investigational Site, Bothell, Washington
  - Otsuka Investigational Site, Richland, Washington
- Argentina (8):
  - Otsuka Investigational Site, Ciudad Autónoma de Bs. As., Buenos Aires
  - Otsuka Investigational Site, La Plata, Buenos Aires
  - Otsuka Investigational Site, Lanús Este, Buenos Aires
  - Otsuka Investigational Site, Córdoba, Córdoba Province
  - Otsuka Investigational Site, Pueyrredón, Córdoba Province
  - Otsuka Investigational Site, Mendoza, Mendoza Province
  - Otsuka Investigational Site, Rosario, Santa Fe Province
  - Otsuka Investigational Site, Buenos Aires
- Bulgaria (8):
  - Otsuka Investigational Site, Lovech
  - Otsuka Investigational Site, Pleven
  - Otsuka Investigational Site, Plovdiv
  - Otsuka Investigational Site, Radnevo
  - Otsuka Investigational Site, Region of Veliko Tarnovo
  - Otsuka Investigational Site, Rousse
  - Otsuka Investigational Site, Sofia
  - Otsuka Investigational Site, Varna
- India (7):
  - Otsuka Investigational Site, Ahmedabad, Gujarat
  - Otsuka Investigational Site, Bangalore, Karnataka
  - Otsuka Investigational Site, Chennai, Tamil Nadu
  - Otsuka Investigational Site, Kanpur
  - Otsuka Investigational Site, Mangalore
  - Otsuka Investigational Site, Pune
  - Otsuka Investigational Site, Tirupati
- Malaysia (4):
  - Otsuka Investigational Site, Cheras, Kuala Lumpur
  - Otsuka Investigational Site, Kuala Lumpur, Kuala Lumpur
  - Otsuka Investigational Site, Tanjong Rambutan, Perak
  - Otsuka Investigational Site, Kuala Selangor
- Mexico (5):
  - Otsuka Investigational Site, Guadalajara, Jalisco
  - Otsuka Investigational Site, Mexico City, Mexico City
  - Otsuka Investigational Site, Monterrey, Nuevo León
  - Otsuka Investigational Site, San Luis Potosí City, San Luis Potosí
  - Otsuka Investigational Site, Culiacán, Sinaloa
- Philippines (5):
  - Otsuka Investigational Site, Bataan, Central Luzon
  - Otsuka Investigational Site, Mandaluyong, NCR
  - Otsuka Investigational Site, Quezon City, NCR
  - Otsuka Investigational Site, Iloilo City, Western Visayas
  - Otsuka Investigational Site, Cebu City
- Romania (6):
  - Otsuka Investigational Site, Arad
  - Otsuka Investigational Site, Bucharest
  - Otsuka Investigational Site, Cluj-Napoca
  - Otsuka Investigational Site, Craiova
  - Otsuka Investigational Site, Oradea
  - Otsuka Investigational Site, Piteşti
- Russia (5):
  - Otsuka Investigational Site, Lipetsk
  - Otsuka Investigational Site, Moscow
  - Otsuka Investigational Site, Nizhny Novgorod
  - Otsuka Investigational Site, Saint Petersburg
  - Otsuka Investigational Site, Smolensk
- Serbia (2):
  - Otsuka Investigational Site, Belgrade
  - Otsuka Investigational Site, Kragujevac
- Slovakia (5):
  - Otsuka Investigational Site, Košice
  - Otsuka Investigational Site, Liptovský Mikuláš
  - Otsuka Investigational Site, Prešov
  - Otsuka Investigational Site, Rimavská Sobota
  - Otsuka Investigational Site, Svidník
- Taiwan (4):
  - Otsuka Investigational Site, Changhua
  - Otsuka Investigational Site, Hualien City
  - Otsuka Investigational Site, Tainan
  - Otsuka Investigational Site, Taipei

REFERENCES:
- [Result] Kane JM, Sanchez R, Perry PP, Jin N, Johnson BR, Forbes RA, McQuade RD, Carson WH, Fleischhacker WW. Aripiprazole intramuscular depot as maintenance treatment in patients with schizophrenia: a 52-week, multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2012 May;73(5):617-24. doi: 10.4088/JCP.11m07530. PMID 22697189
- [Derived] Kane JM, Sanchez R, Baker RA, Eramo A, Peters-Strickland T, Perry PP, Johnson BR, Tsai LF, Carson WH, McQuade RD, Fleischhacker WW. Patient-Centered Outcomes with Aripiprazole Once-Monthly for Maintenance Treatment in Patients with Schizophrenia: Results From Two Multicenter, Randomized, Double-Blind Studies. Clin Schizophr Relat Psychoses. 2015 Summer;9(2):79-87. Epub 2015 Feb 24. PMID 25711509
- [Derived] Fleischhacker WW, Sanchez R, Johnson B, Jin N, Forbes RA, McQuade R, Baker RA, Carson W, Kane JM. Long-term safety and tolerability of aripiprazole once-monthly in maintenance treatment of patients with schizophrenia. Int Clin Psychopharmacol. 2013 Jul;28(4):171-6. doi: 10.1097/YIC.0b013e3283615dba. PMID 23615694

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 4 phases in this study. In phases 1-3 (Conversion Phase, Oral Stabilization Phase, Depot Stabilization Phase), there was a single treatment group. In phase 4 (Depot Maintenance Phase), there were 2 treatment groups. All Outcome Measures were assessed in the Depot Maintenance Phase of the study.
Groups:
- All Patients: During the Conversion Phase, patients were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy. During the Oral Stabilization Phase, patients were stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily. During the Depot Stabilization Phase, patients were stabilized on aripiprazole depot.
Period: Conversion Phase
Arm/Group | All Patients | Aripiprazole Depot | Placebo Depot
Started | 633 | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.)
Received Study Medication | 632 | 0 | 0
Completed | 500 | 0 | 0
Not Completed | 133 | 0 | 0
Not completed — Sponsor Discontinued Study | 54 | 0 | 0
Not completed — Lost to Follow-up | 13 | 0 | 0
Not completed — Met Withdrawal Criteria | 4 | 0 | 0
Not completed — Withdrawn by Investigator | 4 | 0 | 0
Not completed — Withdrew Consent | 24 | 0 | 0
Not completed — Protocol Deviation | 2 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Lack of Efficacy with Adverse Event | 13 | 0 | 0
Not completed — Lack of Efficacy without Adverse Event | 8 | 0 | 0
Period: Oral Stabilization Phase
Arm/Group | All Patients | Aripiprazole Depot | Placebo Depot
Started | 710 (210 of the 710 patients who started this phase enrolled in this study directly into this phase.) | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.)
Received Study Medication | 709 | 0 | 0
Completed | 576 | 0 | 0
Not Completed | 134 | 0 | 0
Not completed — Sponsor Discontinue Study | 42 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0
Not completed — Met Withdrawal Criteria | 19 | 0 | 0
Not completed — Withdrawn by Investigator | 12 | 0 | 0
Not completed — Withdrew Consent | 29 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0
Not completed — Lack of Efficacy with Adverse Event | 7 | 0 | 0
Not completed — Lack of Efficacy without Adverse Event | 4 | 0 | 0
Period: Depot Stabilization Phase
Arm/Group | All Patients | Aripiprazole Depot | Placebo Depot
Started | 576 | 0 (There were no patients in this reporting group in this phase of the study.) | 0 (There were no patients in this reporting group in this phase of the study.)
Completed | 403 | 0 | 0
Not Completed | 173 | 0 | 0
Not completed — Sponsor Discontinued Study | 86 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 0
Not completed — Met Withdrawal Criteria | 8 | 0 | 0
Not completed — Withdrawn by Investigator | 9 | 0 | 0
Not completed — Withdrew Consent | 29 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 0
Not completed — Lack of Efficacy with Adverse Event | 12 | 0 | 0
Not completed — Lack of Efficacy without Adverse Event | 1 | 0 | 0
Period: Depot Maintenance Phase
Arm/Group | All Patients | Aripiprazole Depot | Placebo Depot
Started | 0 (Patients were randomized into the aripiprazole and placebo depot groups in this phase of the study.) | 269 | 134
Completed | 0 | 23 | 3
Not Completed | 0 | 246 | 131
Not completed — Sponsor Discontinued Study | 0 | 179 | 58
Not completed — Lost to Follow-up | 0 | 5 | 3
Not completed — Met Withdrawal Criteria | 0 | 2 | 2
Not completed — Withdrawn by Investigator | 0 | 8 | 6
Not completed — Withdrew Consent | 0 | 14 | 4
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Adverse Event without Impending Relapse | 0 | 9 | 5
Not completed — Impending Relapse with Adverse Event | 0 | 11 | 13
Not completed — Impending Relapse without Adverse Event | 0 | 16 | 40

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the participants from the Depot Maintenance Phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Depot | Placebo Depot | Total
Number analyzed (Participants) | 269 | 134 | 403
Age Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.0) | 41.7 (10.5) | 40.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 55 | 162
  Male | 162 | 79 | 241

OUTCOME MEASURES:

1. Primary Outcome: Time to Exacerbation of Psychotic Symptoms/Impending Relapse
Description: A patient experienced an exacerbation of psychotic symptoms/impending relapse if they met any of the following 4 criteria. 1) Clinical Global Impression of Improvement score ≥ 5 and either an increase on any of the following Positive and Negative Syndrome Scale (PANSS) items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content) to a score > 4 with an increase of ≥ 2 on that item since randomization or an increase on any of the same PANSS items to a score > 4 and an increase of ≥ 4 on the same combined PANSS items since randomization, 2) Hospitalization due to worsening of psychotic symptoms, 3) Clinical Global Impression of Severity of Suicide (CGI-SS) score of 4 or 5 on Part 1 and/or 6 or 7 on Part 2, or 4) Violent behavior resulting in clinically significant self-injury, injury to another person, or property damage.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 269 | 134
Days | NA [NA to NA] — The median and confidence interval were not estimable due to too few events. | 209 [161 to 254]
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Based on 6-month IR rates of 55% for placebo and 35% for aripiprazole, sample sizes were estimated to achieve 90% power to detect a hazard ratio of 0.54 and to preserve an overall nominal alpha level of 0.05 (2-sided), allowing for 2 interim looks at 50% and 75% of events. Assuming that each subject was followed for 12 months after randomization and allowing for a 25% loss to follow-up, the projected total number of subjects to be randomly assigned to treatment in the trial was 225; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.199, 95% CI 2-sided [0.125 to 0.317] — Aripiprazole depot/placebo depot

2. Secondary Outcome: Percentage of Patients Meeting Exacerbation of Psychotic Symptoms/Impending Relapse Criteria
Description: This is the key secondary Outcome Measure.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 269 | 134
Percentage of patients | 10.0 | 39.6
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, Chi-squared — The alpha levels for this key secondary Outcome Measure were the same as used for the primary Outcome Measure

3. Secondary Outcome: Percentage of Responders
Description: A patient was considered to be a responder if all of the following criteria were met. 1) Outpatient status, 2) PANSS total score ≤ 80, 3) Lack of specific psychotic symptoms on the PANSS as measured by a score of ≤ 4 on each of the following items (possible scores of 1 to 7 for each item): Conceptual disorganization, suspiciousness, hallucinatory behavior, unusual thought content, and 4) Clinical Global Impression of Severity of Illness (CGI-S) ≤ 4 (moderately ill) and 5) CGI-SS ≤ 2 (mildly suicidal) on Part 1 and ≤ 5 (minimally worsened) on Part 2.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat (ITT) population: All randomized patients. Two of the 269 patients in the ITT population did not attend the Last Visit at which this Outcome Measure was assessed and were not included in the analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 267 | 134
Percentage of patients | 87.6 | 56.0
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, Chi-squared

4. Secondary Outcome: Percentage of Patients Achieving Remission
Description: A patient was considered to have achieved remission if they had a score of ≤ 3 on each of the following PANSS items, maintained for a period of 6 months: Delusions (P1), unusual thought content (G9), hallucinatory behavior (P3), conceptual disorganization (P2), mannerisms/posturing (G5), blunted affect (N1), social withdrawal (N4), and lack of spontaneity (N6).
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients who stayed in Phase 4 for at least 6 months and had values for the specific PANSS items P1, G9, P3, P2,G5, N1, N4, and N6.
Measure: Number; unit: Percentage of patients
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 87 | 31
Percentage of patients | 52.9 | 38.7
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p = 0.1756, Chi-squared

5. Secondary Outcome: Mean Change From Baseline in the PANSS Total Score
Description: The PANSS consists of 3 subscales (Positive Subscale, 7 constructs, scores ranged from 7-49, Negative Subscale, 7 constructs, scores ranged from 7-49, General Psychopathology Subscale, 16 constructs, scores ranged from 16-112) containing a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. The PANSS total score ranged from 30-210 with a higher score indicating more severe symptoms. A negative change score indicates improvement.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients who had PANSS total scores at both baseline and at least 1 post-baseline time point in Phase 4. Last observation carried forward was implemented to impute the missing data at post-baseline visits. Baseline was not carried forward in imputing the missing data at post-baseline visits.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 25 | 4
Units on a scale | 1.43 (0.756) | 11.55 (1.066)
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA included treatment as a term and baseline as a covariate; Mean Difference (Final Values) = -10.11, 95% CI 2-sided [-12.68 to -7.54]

6. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression - Severity (CGI-S) Score
Description: The severity of illness for each patient was rated using the CGI-S. To assess CGI-S, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The CGI-S score ranged from 0-7 with a higher score indicating greater illness. A negative change score indicates improvement.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients who had CGI-S scores at both baseline and at least 1 post-baseline time point in Phase 4. Last observation carried forward was implemented to impute the missing data at post-baseline visits. Baseline was not carried forward in imputing the missing data at post-baseline visits.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 266 | 134
Units on a scale | 0.14 (0.051) | 0.66 (0.073)
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA included treatment as a term and baseline as a covariate; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.70 to -0.35]

7. Secondary Outcome: Mean Change From Baseline in the PANSS Positive Subscale Score
Description: The PANSS Positive Subscale consists of 7 symptom constructs (delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility). For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Scores on each subscale ranged from 7-49 with a higher score indicating more severe symptoms. A negative change score indicates improvement.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients who had PANSS sub-scale scores at both baseline and at least 1 post-baseline time point in Phase 4. Last observation carried forward was implemented to impute the missing data at post-baseline visits. Baseline was not carried forward in imputing the missing data at post-baseline visits.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 266 | 134
Units on a scale | 0.44 (0.265) | 4.25 (0.374)
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Positive Subscale Score; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA included treatment as a term and baseline as a covariate; Mean Difference (Final Values) = -3.82, 95% CI 2-sided [-4.72 to -2.91]

8. Secondary Outcome: Mean Change From Baseline in the PANSS Negative Subscale Score
Description: The PANSS Negative Subscale consists of 7 symptom constructs (blunted affect, emotional withdrawal, poor rapport, passive pathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking). For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Scores on each subscale ranged from 7-49 with a higher score indicating more severe symptoms. A negative change score indicates improvement.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 266 | 134
Units on a scale | 0.19 (0.201) | 1.55 (0.284)
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p = 0.0001, ANCOVA; The ANCOVA included treatment as a term and baseline as a covariate; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.04 to -0.67]

9. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Score
Description: The efficacy of the study medication was rated for each patient using the CGI-I scale. The rater or investigator rated the patient's total improvement whether or not it was due entirely to drug treatment. All responses were compared to the patient's condition at Baseline. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I score ranged from 0-7 with a higher score indicating less improvement/worsening.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients who had CGI-I scores at both baseline and at least 1 post-baseline time point in Phase 4. Last observation carried forward was implemented to impute the missing data at post-baseline visits. Baseline was not carried forward in imputing the missing data at post-baseline visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 266 | 133
Units on a scale | 3.70 (1.05) | 4.53 (1.23)
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

10. Secondary Outcome: Time to Discontinuation
Description: Time to discontinuation was defined as the date of randomization to the date of study discontinuation.
Time Frame: Baseline of the depot maintenance phase to the end of the study (Week 52)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aripiprazole Depot | Placebo Depot
Number analyzed (Participants) | 269 | 134
Days | NA [364 to NA] — The median and the upper limit of the confidence interval were not estimable due to too few events. | 162 [98 to 211]
Statistical Analysis 1: Comparison: Aripiprazole Depot vs Placebo Depot; Test type: Superiority or Other; p < 0.0001, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the signing of informed consent until the end of the study (up to 106 weeks).
Description: Safety population: All subjects who received at least 1 dose of study medication.
Groups:
- Conversion Phase: During the Conversion Phase, patients were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy.
- Oral Stabilization Phase: During the Oral Stabilization Phase, patients were stabilized on an oral dose of aripiprazole ranging from 10 mg to 30 mg daily.
- Depot Stabilization Phase: During the IM Depot Stabilization Phase, patients were stabilized on aripiprazole IM depot.
- Aripiprazole Depot - Depot Maintenance Phase: Patients received aripiprazole 300 mg or 400 mg depot intramuscularly every 28 days for 52 weeks.
- Placebo Depot - Depot Maintenance Phase: Patients received placebo intramuscularly every 28 days for 52 weeks.
Arm/Group | Conversion Phase | Oral Stabilization Phase | Depot Stabilization Phase | Aripiprazole Depot - Depot Maintenance Phase | Placebo Depot - Depot Maintenance Phase
Serious Adverse Events (participants affected / at risk) | 13/632 | 10/709 | 25/576 | 11/269 | 9/134
Other Adverse Events (participants affected / at risk) | 113/632 | 50/709 | 184/576 | 103/269 | 43/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion Phase (N=632) | Oral Stabilization Phase (N=709) | Depot Stabilization Phase (N=576) | Aripiprazole Depot - Depot Maintenance Phase (N=269) | Placebo Depot - Depot Maintenance Phase (N=134)
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 1 | 2 | 4 | 4
Schizophrenia (Psychiatric disorders) | 6 | 6 | 9 | 2 | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 2 | 1 | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion Phase (N=632) | Oral Stabilization Phase (N=709) | Depot Stabilization Phase (N=576) | Aripiprazole Depot - Depot Maintenance Phase (N=269) | Placebo Depot - Depot Maintenance Phase (N=134)
Headache (Nervous system disorders) | 45 | 23 | 34 | 16 | 7
Insomnia (Psychiatric disorders) | 76 | 50 | 46 | 27 | 12
Injection site pain (General disorders) | 0 | 2 | 34 | 8 | 5
Weight increased (Investigations) | 8 | 16 | 40 | 26 | 13
Akathisia (Nervous system disorders) | 30 | 33 | 36 | 15 | 8
Anxiety (Psychiatric disorders) | 27 | 29 | 38 | 16 | 10
Nasopharyngitis (Infections and infestations) | 14 | 6 | 11 | 10 | 7
Tremor (Nervous system disorders) | 16 | 14 | 21 | 16 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No